CLINICAL TRIAL: NCT04905355
Title: Contribution of Virtual Reality on Patient Satisfaction in Ambulatory Orthopedic Surgery
Brief Title: Virtual Reality on Patient Satisfaction in Ambulatory Orthopedic Surgery
Acronym: SATISVIR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021-A00479-32
Record Dates: First submitted 2021-05-24; First posted 2021-05-27 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Orthopedic
Keywords: Surgery; Virtual Reality; Patient satisfaction; Ambulatory
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Use of VR or not during the ambulatory orthopedic surgery will be attributed to patient randomly.
Who Masked: Outcomes Assessor
Masking Description: Assessor of the main outcome will be not aware of arm attribution
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (VR) (Active Comparator): Patient with VR experience during the ambulatory orthopedic surgery
  Interventions: Device: Virtual reality
- NO VR (No Intervention): Patient without any VR experience during the ambulatory orthopedic surgery

INTERVENTIONS:
Device: Virtual reality — The VR used during the ambulatory orthopedic surgery allows immersive experience in HD-2D virtual environment. Patient can choose among movies, cartoons, entertainments offered for visualization during the surgery
  Arms: Virtual Reality (VR)

SUMMARY:
Few studies were interested in the patient satisfaction after ambulatory surgery. Most of them showed negative results due to psychological factors. The intervention including surgery and hospitalization is still perceived as painful memory for most of patients. Several improving axes have been explored to change global patient experience. One new idea could be to offer a virtual reality experience during the surgery or local regional anesthesia. Some studies showed that immersive experience can reduce the anxiety, the pain, improve the patient comfort and recovery after surgery. The virtual reality is commonly used but it has to be evaluated in terms of efficiency with a prospective study and objective outcomes to go further in the improvement of the experience and the care offer to patients.

DETAILED DESCRIPTION:
The study is to compare the patient satisfaction between patients with virtual reality experience and patients without VR experience during the ambulatory orthopedic surgery under local regional anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Participant who has an ambulatory orthopedic surgery under local regional anesthesia, planned or performed in emergency
* Participant who has been given appropriate information about the study objectives and who has given his/her express written and informed consent prior to conduct any study-related procedures.

Exclusion Criteria:

* Participant with visual deficiency or deaf
* Participant who can bear virtual reality
* Participant whose physical and / or psychological health is severely impaired, which according to the investigator may affect the participant's compliance with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction of operating room management by Net Promoter Score | One Day after surgery
  Net Promoter Score (scale from 0 to 10 with 3 groups: promoters for 9-10, passive for 7-8 and detractor for below 6)

SECONDARY OUTCOMES:
Patient satisfaction of ambulatory hospitalization by e-SATIS questionnaire | One Day after surgery
  e-SATIS questionnaire : measure of hospitalization experience and patient satisfaction (the best scoring is 100 , excellent satisfaction)

OTHER OUTCOMES:
Anesthesia experience by EVAN-LR questionnaire | One Day after surgery
  EVAN-LR (Evaluation du Vécu de l'ANesthésie - Local Regionale) questionnaire: five-point Likert scale, defined from 1 to 5 as "much less than expected," "less than expected," "as expected," "more than expected," and "much more than expected." All dimension scores are linearly transformed to a 0-100 scale, with 100 indicating the best possible level of satisfaction and 0 the worst.
Functional outcomes by measurement of symptoms as well as the ability to perform certain activities. (QUICKDASH questionnaire) | One month after surgery
  Quick DASH( Disabilities of the Arm, Shoulder and Hand) questionnaire : 11 items with 5 response options. Scale scores are calculated ranging from 0 (no disability) to 100 (more severe disability)

CONTACTS AND LOCATIONS:
Locations (1):
- RGDS-Clinique Aguiléra, Biarritz, France

IPD SHARING:
Plan to Share IPD: No